CLINICAL TRIAL: NCT06611228
Title: Optimizing Prevention of Hospital-acquired Disability Through Integrated Multidomain Interventions: the Age-IT Project
Brief Title: Optimizing Prevention of Hospital-Acquired Disability Through Multidomain Interventions
Acronym: OPTIMAge-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OPTIMAge-IT
Record Dates: First submitted 2024-09-02; First posted 2024-09-24 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-11

CONDITIONS: Frailty Syndrome; Aging
Keywords: Hospital Acquired Disability; Frailty Syndrome; Comprehensive Geriatric Assessment; Prevention; Integrated Multidomain Interventions; Telemedicine; Telemonitoring; Outcomes; Hospital
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Pragmatic, randomized controlled (parallel-arm cluster), non-drug interventional clinical study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The interventions include:
  * Physical Exercise: Tailored sessions with the VIVIFRAIL exercise protocol, monitored with accelerometers, and supported by a physical activity kit.
  * Nutrition: Mediterranean diet with education on nutrient balance and avoiding ultra-processed foods.
  * Health & Sleep: Promotion of healthy habits, fall prevention, sleep hygiene, and targeted sleep disorder treatments.
  * Polypharmacotherapy: Review and adjustment of medications as needed.
  * Cognition: Cognitive rehabilitation using technology and educational videos.
  * Environment: Adjustments to create an "older-friendly" Acute Unit, including modified routines and extended visiting hours.
  Interventions: Other: Multidomain Interventions
- Control Group (No Intervention): Centers randomized to the control group will follow usual care protocols. However, all participants in this group will receive standardized leaflets at discharge, providing physical, nutritional, and behavioral advice.

INTERVENTIONS:
Other: Multidomain Interventions — Multidomain Interventions The intervention group will receive a personalized MDI approach from a multidisciplinary team, including a digital coach, physiotherapist, clinical nutrition expert, neuropsychologist, geriatrician, and nurse. This approach will encompass physical activity program, nutritional interventions, cognitive training and stimulation, medication reconciliation, coaching on the use of technological supports, and group activities. Environmental modifications at home will also be proposed
  Arms: Intervention Group

SUMMARY:
The aim of this study is to assess whether a multidomain, multidisciplinary intervention (MDI), enhanced by technological solutions, effectively improves the functional and cognitive status of older hospitalized patients at risk of disability or worsening frailty. Additionally, the study will evaluate the feasibility and acceptability of delivering these interventions remotely via technology after hospital discharge.

Participants will:

* Receive an MDI during their hospital stay and continue with remote at-home support for 3 months, or receive usual care.
* Attend outpatient clinics for follow-up assessment at 3 and 6 months.

DETAILED DESCRIPTION:
The "Optimizing Prevention of Hospital-Acquired Disability Through Integrated Multidomain Interventions (OPTIMAge-IT)" study will evaluate impact of a MDI multidisciplinary approach, enhanced by technological solutions, on the functional and cognitive status of older hospitalized patients at risk of disability or worsening frailty.

Additionally, the study will evaluate the feasibility and acceptability of delivering MDIs remotely via technology after hospital discharge. Using a parallel cluster-randomized design, approximately 300 patients will be recruited from eight Acute Geriatric Units (AGUs) located in eight acute hospitals evenly distributed across Northern, Central, and Southern Italy.

Eligible patients will be aged 70 years or older, with mild to moderate frailty, capable of ambulation with or without assistance and able to communicate and collaborate with the research team. Participants will use smart technologies, such as smartwatches, and tablets, for guided physical activity and remote monitoring. A multidisciplinary team -including a geriatrician, a nurse, a physiotherapist, a clinical nutrition expert, a neuropsychologist and a digital coach- will assist patients in the intervention group, supervising the MDI approach during hospitalization and at the 3-month follow-up. Blood-based biomarkers and fecal samples for gut microbiome analysis will be collected for patients in the intervention group, to support frailty stratification at baseline and help define the trajectories of functional and cognitive changes from baseline to follow-up assessments.

After discharge, patients in the intervention group will continue MDI at home for 12 weeks, with follow-up visits at 3 and 6 months. The control group will receive a follow-up visit at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >70 years;
* Mild to moderate frailty, defined by a panel of tools agreed upon by the group of researchers involved in the study (Primary Care Frailty Index [PC-FI] between 0.07 and 0.21, Clinical Frailty Scale [CFS] 4-6);
* Ability to walk with or without assistance
* Ability to communicate and cooperate with the research team;
* Ability to sign informed consent.

Exclusion Criteria:

* Expected hospital stay duration <3 days;
* Estimated prognosis quoad vitam <12 months;
* Persistent clinical instability, indicated by a NEWS2 score >5 (assessed within 48 hours of admission) and/or the presence of delirium (4AT >4);
* History of schizophrenia, major depression, bipolar disorder, or psychosis;
* Severe sensory deficits (visual and auditory);
* Presence of a nasogastric tube or percutaneous endoscopic gastrostomy (PEG);
* Severe cardiac conduction disorder (e.g., third-degree atrioventricular block), uncontrolled arrhythmia, new Q wave in the past six months, or ST segment depression (>3 mm) on the electrocardiogram;
* Terminal stage oncological or organic disease (e.g., Child-Pugh C cirrhosis, stage V renal disease, GOLD stage D chronic obstructive pulmonary disease, end-stage heart failure);
* Residence in a nursing home before hospital admission;
* Presence of dissected aortic aneurysm, severe aortic stenosis, acute endocarditis/pericarditis, acute thromboembolism, uncontrolled hypertension (>180/100 mmHg) or postural hypotension, uncontrolled hypoglycemia, recent fracture within the last month, or any other medical condition that hinders the execution of physical activity according to clinical judgment;
* Any condition that prevents safe participation in the intervention and/or cooperation with the study;
* Concurrent participation in other clinical studies;
* Clinical conditions or situations significantly different from the condition under study, which in the investigator's opinion could interfere with the study or prevent optimal participation;
* Participants refusal to participate in the study.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the feasibility of home-based MDI with technological support | 3 months, and 6 months
  Feasibility of home-based MDI with technological support, evaluated using Patient Reported Experience Measures (PREMs), questionnaires measuring the patients' perceptions of their experience whilst receiving care
Evaluate the participant adherence to the protocol | through study completion, an average of 1 year
  Evaluate the participant adherence to the protocol assessing the number of drop-out and overall retention rates
Assess the effect of the MDI on motor function at discharge from the AGU | Baseline, Discharge (after an average hospital stay of 10 days)
  Effect of the intervention in terms of motor function, assessed using the Short Physical Performance Battery (SPPB, from 0 to 12)

SECONDARY OUTCOMES:
Assess the effect of the MDI on readmissions at 6 months follow-up. | 6 months
  Effect of the MDI in reducing hospital readmissions at 6 months
Assess the effect of the MDI on readmissions at 3 months follow-up. | 3 months
  Effect of the MDI in reducing hospital readmissions at 3 months
Evaluate the effect of the MDI on quality of life at follow-up. | 3 months, 6 months
  Effect of the MDI on participants' quality of life at follow-up, evaluated using the EuroQol EQ-5D 5L, a descriptive system comprising five dimensions (mobility, self-care, usual activities, discomfort, and anxiety/depression), each dimension with five response levels (no problems, slight problems, moderate problems, severe problems, unable to/extreme problems).
Evaluate the effect of the MDI on in-hospital mortality | From Admission Through Discharge, an Average of 10 days
  Evaluate the effect of the MDI on in-hospital mortality
Evaluate the effect of the MDI on mortality at follow-up. | 3 months, 6 months
  Evaluate the effect of the MDI on mortality at follow-up.
Evaluate the effect of the MDI on dietary intake and nutritional status at follow-up. | Baseline, 3 months, 6 months
  Effect of the MDI in improving dietary intake and nutritional status at follow-up, assessed using the Mediterranean Diet Scale (MDScale, that includes nine components) and Mini Nutritional Assessment-Short Form (MNA-SF, 0-14)
Evaluate the effect of the MDI on changes in frailty levels at follow-up. | Baseline, 3 months, 6 months
  Effect of the MDI in reducing frailty at follow-up, assessed using the Clinical Frailty Scale (CFS, 0-9) and Primary Care Frailty Index (PC-FI)
Assess the effect of the MDI on fall events | Baseline, From Admission Through Discharge, an Average of 10 days, 3 months, 6 months
  Effect of the MDI in reducing the incidence of falls during hospitalization and at home, evaluated through the number of falls and the Tinetti Scale (0-28) occurred within the study period
Evaluate the effect of the MDI on in-hospital complications | Baseline, From Admission Through Discharge, an Average of 10 days, 3 months, 6 months
  Effect of the MDI in reducing the incidence of in-hospital complications as sepsis, urinary infections, blood infections, and pressure ulcers.
Assess the effect of the MDI on sleep quality | Baseline, From Admission Through Discharge, an Average of 10 days, 3 months, 6 months
  Effect of the MDI on sleep quality during hospitalization and at home, assessed using the Pittsburgh Sleep Quality Index (PSQI). The questionnaire consists of a combination of Likert-type and open-ended questions (which can later be converted into scaled scores using appropriate guidelines).
Assess the effect of the MDI on the incidence of delirium during hospitalization | From Admission Through Discharge, an Average of 10 days
  Effect of the MDI in reducing incident delirium during hospitalization, diagnosed according to international guidelines (DSM V) and assessed using the Modified Richmond Agitation Screening Scale (m-RASS, scoring from -5 to +4), 4AT (scoring, from 0 to 12), and Delirium Rating Scale (DRS-revised, 13 items, each item is rated on a scale of 0- 2/3)
Assess the effect of the MDI on cognitive performance at follow-up. | Baseline, From Admission Through Discharge, an Average of 10 days, 3 months, 6 months
  Effect of the MDI on cognitive performance (assessed using the Cognitive Reserve Index questionnaire (CRIq), Addenbrooke Cognitive Examination - Revised (ACE-R), Trail Making Test (TMT) parts A and B)
Assess the effect of the MDI on functional performance at follow-up | Baseline, From Admission Through Discharge, an Average of 10 days, 3 months, 6 months
  Assessed using Basic Activities of Daily Living (ADL 0-6), Instrumental Activities of Daily Living (IADL 0-8), Barthel Index at follow-up (0-100)
Assess the effect of the MDI on motor performance at follow-up. | Baseline, From Admission Through Discharge, an Average of 10 days, 3 months, 6 months
  Assessed using SPPB (0-12), hand grip strength (Kg)
Assess the acceptability of technological solutions during hospitalization and at follow-up. | Discharge (after an average hospital stay of 10 days), 3 months, and 6 months
  Acceptability of technological solutions through the administration of specific questionnaires
Evaluate the cost impact of the MDI on the healthcare system. | Discharge (after an average hospital stay of 10 days), 3 months, and 6 months
  Costs of the MDI on the healthcare system, evaluated through the incremental cost-effectiveness ratio
Evaluate the effect of the MDI on the length of hospital stay. | Discharge (after an average hospital stay of 10 days)
  Effect of the MDI in reducing the length of hospital stay

OTHER OUTCOMES:
Assess the impact of the MDI on cardiovascular risk factors. | Baseline, 6 months
  Impact of MDI on lifestyle and inactivity, blood pressure, smoking, cholesterol level, and blood glucose.
Evaluate the effect of the MDI on participants&amp;#39; social relationships. | 3 months, 6 months
  Effect of the MDI on improving social relationships, assessed using the Lubben Social Network Scale (12 items scale)
Evaluate the impact of fortified food consumption on microbiota composition and bowel alterations in a subgroup of patients not undergoing antibiotic therapy (ancillary study). | Baseline, Through Discharge an Average of 10 days
  Evaluation of the impact of fortified food consumption on faecal analysis in a subgroup of patients not undergoing antibiotic therapy
Assess participants access to (and frequency of use of) technological resources. | Through Discharge an Average of 10 days, 3 months
  Number of app accesses.
Assess the effect of the MDI on mood of participants | Baseline, 3 months, 6 months
  Effect of the MDI on mood, assessed using the Geriatric Depression Scale (GDS, 0-30)
Evaluate the effect of the MDI on biomarkers of aging | Baseline, 6 months
  Changes on the Free Triiodothyronine/Free Thyroxine (FT3/FT4) concentration in the MDI group compared to controls
Evaluate the effect of the MDI on biomarkers of aging | Baseline
  Effect of the MDI on partipants according to Serum Amyloid Beta (Aβ) concentration categories
Evaluate the effect of the MDI on biomarkers of aging | Baseline
  Effect of the MDI on partipants according to their Serum Phosphorylated Tau at Threonine 181 (p-tau181), p-tau217, p-tau231 concentrations
Evaluate the effect of the MDI on biomarkers of aging | Baseline, 6 months
  Changes on high-sensitivity C-reactive protein (hs-CRP, measured in mg/L) concentration of the MDI group compared to controls
Evaluate the effect of the MDI on biomarkers of aging | Baseline, 6 months
  Changes on Erythrocyte sedimentation rate (ESR, measured in mm/h) of the MDI group compared to controls
Evaluate the effect of the MDI on biomarkers of aging | Baseline, 6 months
  Changes on interleukin 6 (IL-6, measured in pg/mL) concentration of the MDI group compared to controls
Evaluate the effect of the MDI on biomarkers of aging | Baseline, 6 months
  Changes on the Neurofilament Light Chain (NF-L, measured in pg/mL) concentration in the MDI group compared to controls
Evaluate the effect of the MDI on biomarkers of aging | Baseline, 6 months
  Changes on the Soluble Receptor for Advanced Glycation End-products (s-RAGE, measured in ng/mL) concentration in the MDI group compared to controls
Evaluate the effect of the MDI on biomarkers of aging | Baseline, 6 months
  Changes on the Fibroblast Growth Factor 1 concentration (FGF-1, measured in pg/mL) in the MDI group compared to controls
Evaluate the effect of the MDI on biomarkers of aging | Baseline, 6 months
  Changes on the Growth Differentiation Factor 15 concentration (GDF-15, measured in pg/mL), in the MDI group compared to controls.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Bellelli, MD, Principal Investigator — Università di Milano-Bicocca; Giuseppe Bellelli, MD, Study Chair — Università di Milano-Bicocca
Locations (1):
- Fondazione IRCCS San Gerardo dei Tintori, Monza, Lumbardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Belloni G, Cesari M. Frailty and Intrinsic Capacity: Two Distinct but Related Constructs. Front Med (Lausanne). 2019 Jun 18;6:133. doi: 10.3389/fmed.2019.00133. eCollection 2019. PMID 31275941
- [Background] Dent E, Martin FC, Bergman H, Woo J, Romero-Ortuno R, Walston JD. Management of frailty: opportunities, challenges, and future directions. Lancet. 2019 Oct 12;394(10206):1376-1386. doi: 10.1016/S0140-6736(19)31785-4. PMID 31609229
- [Background] Thillainadesan J, Scott IA, Le Couteur DG. Frailty, a multisystem ageing syndrome. Age Ageing. 2020 Aug 24;49(5):758-763. doi: 10.1093/ageing/afaa112. PMID 32542377
- [Background] Lee H, Lee E, Jang IY. Frailty and Comprehensive Geriatric Assessment. J Korean Med Sci. 2020 Jan 20;35(3):e16. doi: 10.3346/jkms.2020.35.e16. PMID 31950775
- [Background] Dedeyne L, Deschodt M, Verschueren S, Tournoy J, Gielen E. Effects of multi-domain interventions in (pre)frail elderly on frailty, functional, and cognitive status: a systematic review. Clin Interv Aging. 2017 May 24;12:873-896. doi: 10.2147/CIA.S130794. eCollection 2017. PMID 28579766
- [Background] de Souto Barreto P, Rolland Y, Maltais M, Vellas B; MAPT Study Group. Associations of Multidomain Lifestyle Intervention with Frailty: Secondary Analysis of a Randomized Controlled Trial. Am J Med. 2018 Nov;131(11):1382.e7-1382.e13. doi: 10.1016/j.amjmed.2018.06.002. Epub 2018 Jul 1. PMID 29969614
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Background] Ellis G, Gardner M, Tsiachristas A, Langhorne P, Burke O, Harwood RH, Conroy SP, Kircher T, Somme D, Saltvedt I, Wald H, O'Neill D, Robinson D, Shepperd S. Comprehensive geriatric assessment for older adults admitted to hospital. Cochrane Database Syst Rev. 2017 Sep 12;9(9):CD006211. doi: 10.1002/14651858.CD006211.pub3. PMID 28898390
- [Background] Ferrara MC, Perez LM, Sole AR, Villa-Garcia L, Ars J, Soto-Bagaria L, Bellelli G, Cesari M, Enfedaque MB, Inzitari M. Sustained improvement of intrinsic capacity in community-dwelling older adults: The +AGIL Barcelona multidomain program. J Intern Med. 2023 Dec;294(6):730-742. doi: 10.1111/joim.13710. Epub 2023 Aug 21. PMID 37574781
- [Background] Kivipelto M, Mangialasche F, Ngandu T. Lifestyle interventions to prevent cognitive impairment, dementia and Alzheimer disease. Nat Rev Neurol. 2018 Nov;14(11):653-666. doi: 10.1038/s41582-018-0070-3. PMID 30291317
- [Background] Perez LM, Enfedaque-Montes MB, Cesari M, Soto-Bagaria L, Gual N, Burbano MP, Tarazona-Santabalbina FJ, Casas RM, Diaz F, Martin E, Gomez A, Orfila F, Inzitari M. A Community Program of Integrated Care for Frail Older Adults: +AGIL Barcelona. J Nutr Health Aging. 2019;23(8):710-716. doi: 10.1007/s12603-019-1244-4. PMID 31560028
- [Background] Casas-Herrero A, Saez de Asteasu ML, Anton-Rodrigo I, Sanchez-Sanchez JL, Montero-Odasso M, Marin-Epelde I, Ramon-Espinoza F, Zambom-Ferraresi F, Petidier-Torregrosa R, Elexpuru-Estomba J, Alvarez-Bustos A, Galbete A, Martinez-Velilla N, Izquierdo M. Effects of Vivifrail multicomponent intervention on functional capacity: a multicentre, randomized controlled trial. J Cachexia Sarcopenia Muscle. 2022 Apr;13(2):884-893. doi: 10.1002/jcsm.12925. Epub 2022 Feb 11. PMID 35150086
- [Background] Courel-Ibanez J, Buendia-Romero A, Pallares JG, Garcia-Conesa S, Martinez-Cava A, Izquierdo M. Impact of Tailored Multicomponent Exercise for Preventing Weakness and Falls on Nursing Home Residents' Functional Capacity. J Am Med Dir Assoc. 2022 Jan;23(1):98-104.e3. doi: 10.1016/j.jamda.2021.05.037. Epub 2021 Jun 29. PMID 34197791
- [Background] Martinez-Velilla N, Casas-Herrero A, Zambom-Ferraresi F, Saez de Asteasu ML, Lucia A, Galbete A, Garcia-Baztan A, Alonso-Renedo J, Gonzalez-Glaria B, Gonzalo-Lazaro M, Apezteguia Iraizoz I, Gutierrez-Valencia M, Rodriguez-Manas L, Izquierdo M. Effect of Exercise Intervention on Functional Decline in Very Elderly Patients During Acute Hospitalization: A Randomized Clinical Trial. JAMA Intern Med. 2019 Jan 1;179(1):28-36. doi: 10.1001/jamainternmed.2018.4869. PMID 30419096
- [Background] Creditor MC. Hazards of hospitalization of the elderly. Ann Intern Med. 1993 Feb 1;118(3):219-23. doi: 10.7326/0003-4819-118-3-199302010-00011. PMID 8417639
- [Background] Covinsky KE, Pierluissi E, Johnston CB. Hospitalization-associated disability: "She was probably able to ambulate, but I'm not sure". JAMA. 2011 Oct 26;306(16):1782-93. doi: 10.1001/jama.2011.1556. PMID 22028354
- [Background] Loyd C, Markland AD, Zhang Y, Fowler M, Harper S, Wright NC, Carter CS, Buford TW, Smith CH, Kennedy R, Brown CJ. Prevalence of Hospital-Associated Disability in Older Adults: A Meta-analysis. J Am Med Dir Assoc. 2020 Apr;21(4):455-461.e5. doi: 10.1016/j.jamda.2019.09.015. Epub 2019 Nov 14. PMID 31734122
- [Background] Reichardt LA, Aarden JJ, van Seben R, van der Schaaf M, Engelbert RH, Bosch JA, Buurman BM; Hospital-ADL study group. Unravelling the potential mechanisms behind hospitalization-associated disability in older patients; the Hospital-Associated Disability and impact on daily Life (Hospital-ADL) cohort study protocol. BMC Geriatr. 2016 Mar 5;16:59. doi: 10.1186/s12877-016-0232-3. PMID 26945587
- [Background] Hshieh TT, Inouye SK, Oh ES. Delirium in the Elderly. Psychiatr Clin North Am. 2018 Mar;41(1):1-17. doi: 10.1016/j.psc.2017.10.001. Epub 2017 Dec 22. PMID 29412839
- [Background] Bellelli G, Nobili A, Annoni G, Morandi A, Djade CD, Meagher DJ, Maclullich AM, Davis D, Mazzone A, Tettamanti M, Mannucci PM; REPOSI (REgistro POliterapie SIMI) Investigators. Under-detection of delirium and impact of neurocognitive deficits on in-hospital mortality among acute geriatric and medical wards. Eur J Intern Med. 2015 Nov;26(9):696-704. doi: 10.1016/j.ejim.2015.08.006. Epub 2015 Aug 31. PMID 26333532
- [Background] Fortinsky RH, Covinsky KE, Palmer RM, Landefeld CS. Effects of functional status changes before and during hospitalization on nursing home admission of older adults. J Gerontol A Biol Sci Med Sci. 1999 Oct;54(10):M521-6. doi: 10.1093/gerona/54.10.m521. PMID 10568535
- [Background] Sager MA, Franke T, Inouye SK, Landefeld CS, Morgan TM, Rudberg MA, Sebens H, Winograd CH. Functional outcomes of acute medical illness and hospitalization in older persons. Arch Intern Med. 1996 Mar 25;156(6):645-52. PMID 8629876
- [Background] Sager MA, Rudberg MA, Jalaluddin M, Franke T, Inouye SK, Landefeld CS, Siebens H, Winograd CH. Hospital admission risk profile (HARP): identifying older patients at risk for functional decline following acute medical illness and hospitalization. J Am Geriatr Soc. 1996 Mar;44(3):251-7. doi: 10.1111/j.1532-5415.1996.tb00910.x. PMID 8600192
- [Background] Bellelli G, Morandi A, Di Santo SG, Mazzone A, Cherubini A, Mossello E, Bo M, Bianchetti A, Rozzini R, Zanetti E, Musicco M, Ferrari A, Ferrara N, Trabucchi M; Italian Study Group on Delirium (ISGoD). "Delirium Day": a nationwide point prevalence study of delirium in older hospitalized patients using an easy standardized diagnostic tool. BMC Med. 2016 Jul 18;14:106. doi: 10.1186/s12916-016-0649-8. PMID 27430902
- [Background] Lipowski ZJ. Transient cognitive disorders (delirium, acute confusional states) in the elderly. Am J Psychiatry. 1983 Nov;140(11):1426-36. doi: 10.1176/ajp.140.11.1426. PMID 6624987
- [Background] Lindroth H, Bratzke L, Purvis S, Brown R, Coburn M, Mrkobrada M, Chan MTV, Davis DHJ, Pandharipande P, Carlsson CM, Sanders RD. Systematic review of prediction models for delirium in the older adult inpatient. BMJ Open. 2018 Apr 28;8(4):e019223. doi: 10.1136/bmjopen-2017-019223. PMID 29705752
- [Background] Bellelli G, Mazzone A, Morandi A, Latronico N, Perego S, Zazzetta S, Mazzola P, Annoni G. The Effect of an Impaired Arousal on Short- and Long-Term Mortality of Elderly Patients Admitted to an Acute Geriatric Unit. J Am Med Dir Assoc. 2016 Mar 1;17(3):214-9. doi: 10.1016/j.jamda.2015.10.002. Epub 2015 Nov 12. PMID 26585091
- [Background] Geyskens L, Jeuris A, Deschodt M, Van Grootven B, Gielen E, Flamaing J. Patient-related risk factors for in-hospital functional decline in older adults: A systematic review and meta-analysis. Age Ageing. 2022 Feb 2;51(2):afac007. doi: 10.1093/ageing/afac007. PMID 35165688
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Fisher S, Ottenbacher KJ, Goodwin JS, Graham JE, Ostir GV. Short Physical Performance Battery in hospitalized older adults. Aging Clin Exp Res. 2009 Dec;21(6):445-52. doi: 10.1007/BF03327444. PMID 20154514
- [Background] Guralnik JM, Ferrucci L, Simonsick EM, Salive ME, Wallace RB. Lower-extremity function in persons over the age of 70 years as a predictor of subsequent disability. N Engl J Med. 1995 Mar 2;332(9):556-61. doi: 10.1056/NEJM199503023320902. PMID 7838189
- [Background] Penninx BW, Ferrucci L, Leveille SG, Rantanen T, Pahor M, Guralnik JM. Lower extremity performance in nondisabled older persons as a predictor of subsequent hospitalization. J Gerontol A Biol Sci Med Sci. 2000 Nov;55(11):M691-7. doi: 10.1093/gerona/55.11.m691. PMID 11078100
- [Background] Miller DK, Wolinsky FD, Andresen EM, Malmstrom TK, Miller JP. Adverse outcomes and correlates of change in the Short Physical Performance Battery over 36 months in the African American health project. J Gerontol A Biol Sci Med Sci. 2008 May;63(5):487-94. doi: 10.1093/gerona/63.5.487. PMID 18511752
- [Background] Pavasini R, Guralnik J, Brown JC, di Bari M, Cesari M, Landi F, Vaes B, Legrand D, Verghese J, Wang C, Stenholm S, Ferrucci L, Lai JC, Bartes AA, Espaulella J, Ferrer M, Lim JY, Ensrud KE, Cawthon P, Turusheva A, Frolova E, Rolland Y, Lauwers V, Corsonello A, Kirk GD, Ferrari R, Volpato S, Campo G. Short Physical Performance Battery and all-cause mortality: systematic review and meta-analysis. BMC Med. 2016 Dec 22;14(1):215. doi: 10.1186/s12916-016-0763-7. PMID 28003033
- [Background] Cooper R, Kuh D, Cooper C, Gale CR, Lawlor DA, Matthews F, Hardy R; FALCon and HALCyon Study Teams. Objective measures of physical capability and subsequent health: a systematic review. Age Ageing. 2011 Jan;40(1):14-23. doi: 10.1093/ageing/afq117. Epub 2010 Sep 15. PMID 20843964
- [Background] Bellelli G, Morandi A, Davis DH, Mazzola P, Turco R, Gentile S, Ryan T, Cash H, Guerini F, Torpilliesi T, Del Santo F, Trabucchi M, Annoni G, MacLullich AM. Validation of the 4AT, a new instrument for rapid delirium screening: a study in 234 hospitalised older people. Age Ageing. 2014 Jul;43(4):496-502. doi: 10.1093/ageing/afu021. Epub 2014 Mar 2. PMID 24590568
- See also: Organization WH. World report on ageing and health [Internet]. Geneva PP - Geneva: World Health Organization — https://apps.who.int/iris/handle/10665/186463
- See also: Organization WH. Integrated care for older people: guidelines on community-level interventions to manage declines in intrinsic capacity [Internet]. Geneva PP - Geneva: World Health Organization; — https://apps.who.int/iris/handle/10665/258981